CLINICAL TRIAL: NCT03008005
Title: Effects of THC on Retention of Memory for Fear Extinction Learning in PTSD: R61 Study
Brief Title: Effects of Delta-9 Tetrahydrocannabinol (THC) on Retention of Memory for Fear Extinction Learning in PTSD: R61 Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Christine Rabinak, PhD, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R61MH111935-01 (NIH)
Record Dates: First submitted 2016-12-23; First posted 2017-01-02 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: PostTraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sugars; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Oral Capsule (Placebo Comparator): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (5mg or 10mg) or placebo (PBO) approximately two hours prior to MR scanning and task performance in 78 patients with PTSD.
  One-third of the participants will receive 5mg dronabinol (n=26) , one-third of the participants will receive 10mg dronabinol (n=26), and the remaining one-third of the participants will receive placebo (n=26).
  Interventions: Drug: Placebo Oral Capsule
- Dronabinol Cap 5 milligrams (MG) (Experimental): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (5mg or 10mg) or placebo (PBO) approximately two hours prior to MR scanning and task performance in 78 patients with PTSD.
  One-third of the participants will receive 5mg dronabinol (n=26) , one-third of the participants will receive 10mg dronabinol (n=26), and the remaining one-third of the participants will receive placebo (n=26).
  Interventions: Drug: Dronabinol Cap 5 milligrams (MG)
- Dronabinol Cap 10 milligrams (MG) (Experimental): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (5mg or 10mg) or placebo (PBO) approximately two hours prior to MR scanning and task performance in 78 patients with PTSD.
  One-third of the participants will receive 5mg dronabinol (n=26) , one-third of the participants will receive 10mg dronabinol (n=26), and the remaining one-third of the participants will receive placebo (n=26).
  Interventions: Drug: Dronabinol Cap 10 milligrams (MG)

INTERVENTIONS:
Drug: Placebo Oral Capsule — Placebo is administered only once (approximately 120 min prior to MR scanning in Visit 3) by the oral route and contains only dextrose in opaque capsules.
  Other Names: sugar pill
  Arms: Placebo Oral Capsule
Drug: Dronabinol Cap 5 milligrams (MG) — Dronabinol (5mg) is administered only once (approximately 120 min prior to MR scanning in Visit 3) by the oral route and is placed in an opaque capsule with dextrose filler.
  Other Names: Marinol
  Arms: Dronabinol Cap 5 milligrams (MG)
Drug: Dronabinol Cap 10 milligrams (MG) — Dronabinol (10mg) is administered only once (approximately 120 min prior to MR scanning in Visit 3) by the oral route and is placed in an opaque capsule with dextrose filler.
  Other Names: Marinol
  Arms: Dronabinol Cap 10 milligrams (MG)

SUMMARY:
The goal of this study is to look at how a type of drug called cannabinoids are related to the processing of fear signals, the experience of emotions and fear, and the pattern of activity in the brain that is involved in these processes and how this relates to the development of post-traumatic stress disorder (PTSD). PTSD is an anxiety disorder that occurs after experiencing a traumatic event(s) and is characterized by unwanted memories of the trauma(s) through flashbacks or nightmares, avoidance of situations that remind the person of the event, difficulty experiencing emotions, loss of interest in activities the person used to enjoy, and increased arousal, such as difficulty falling asleep or staying asleep, anger and hypervigilance. The information gained from this study could lead to the development of new treatments for persons who suffer from anxiety or fear-based disorders.

DETAILED DESCRIPTION:
The total time that for each participant involved in this study is 5 visits, as outlined below:

Visit 1: Questionnaires, Screening, and Orientation: During this visit the potential participant will learn about the study procedures, sign the informed consent documents, and fill out a packet of forms that ask about his or her race and ethnic background, use of drugs and alcohol and physical and mental health.

Visit 2: Behavioral Tests: During this visit the participant will complete several computer tasks, and the study staff will be measuring reaction time and psychophysiological measures.The tasks that the participant will perform will show three different images and an aversive stimulus (e.g. loud burst of noise or animated snake) may follow one image most of the time, while the other images may never be followed by the aversive cue. The participant will need to try to predict whether the aversive cue will occur or not based on which image is shown and will be asked to repeatedly rate on a scale how likely it is that he or she thinks an aversive cue will occur after each image. Lastly, during the session the participant will also be asked to report his or her level of anxiety on a scale from 0 to 100.

Visit 3: Behavioral Tests with Drug or Placebo and Magnetic Resonance (MR) scan: For safety reasons participant will not be allowed to take any drugs for at least 24 hours before this visit, and should not use marijuana for at least 2 weeks before. Participants will be required to pass a urine drug test (and pregnancy test for women) and breathalyzer test before being allowed to continue with this visit. The participant will also not be allowed to drive himself or herself home from this visit, so he or she should arrange a friend or family member to pick him or her up or a taxi can be called by our research staff.

The participant will view the same images he or she did on the previous day (Visit 2), and may experience the same aversive stimulus as during Visit 2. The participant will again be asked to rate how much he or she expects to experience the aversive stimulus after each image and he or she will also be asked to report his or her level of anxiety on a scale from 0 to 100. However, about 2 hours before the task begins, the participant will be asked to swallow a capsule containing either a marijuana-like drug (Dronabinol) or a placebo (sugar pill). Dronabinol is a Food & Drug Administration (FDA) approved drug and the doses (5mg or 10mg; one time) are unlikely to have any effects that last beyond the duration of the study visit. About every 30 minutes after taking the pill, the participant will fill out some questionnaires about mood and how he or she is feeling at the moment.

Visit 4: Behavioral Tests and MR scan: This visit will be very similar to Visit 2. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will view the same images he or she did previously, and may experience the same aversive stimulus as during Visit 2. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

Visit 5: Behavioral Tests and MR scan: This visit will occur approximately 1 week after Visit 4 and will have the same procedure. Participants will participate in the same type of task inside the MR scanner, while the study staff measures reaction time and psychophysiological responding and brain activation. Participants will again be asked to rate how much they expect to experience the aversive stimulus after each image and will also be asked to report their level of anxiety on a scale from 0 to 100.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Right-handed
* Age between 18-50 years old,
* Physically and neurologically healthy [confirmed by a comprehensive medical history]
* Current PTSD diagnosis

Exclusion Criteria:

* clinically significant medical or neurologic condition or neurocognitive dysfunction that would affect function and/or task performance and/or interfere with the study protocol
* any current (or within past 2 months) medical condition requiring medication that would interact with dronabinol or interfere with the study protocol
* risk of harm to self or others that requires immediate intervention
* presence of contraindications, current or past allergic or adverse reaction, or known sensitivity to cannabinoid-like substances (dronabinol/marijuana/cannabis/THC, cannabinoid oil, sesame oil, gelatin, glycerin, and titanium dioxide)
* lack of fluency in English
* positive drug screen or alcohol breathalyzer
* unwilling/unable to sign informed consent document
* currently pregnant (positive pregnancy test), planning pregnancy, or lactating (women)
* under 18 or over 50 years of age
* traumatic brain injury (as defined by The American Congress of Rehabilitation as a person who has had a traumatically induced physiological disruption of brain function (i.e., the head being struck, the head striking an object, and/or the brain undergoing an acceleration/deceleration movement (i.e., whiplash) without direct external trauma to the head), as manifested by at least one of the following: any loss of consciousness; any loss of memory for events immediately before or after the injury; any alteration in mental status at the time of the incident; or focal neurological deficits that may or may not be transient)
* inability to tolerate small, enclosed spaces without anxiety (e.g. claustrophobia), as determined by self-report and/or a preliminary session in a mock scanner
* left-handed;
* presence of ferrous-containing metals within the body (e.g., aneurysm clips, shrapnel/retained particles)
* anticipation of a required drug test in the 4 weeks following the study.
* current diagnosis of a mood, anxiety, or other disorder that is more clinically salient than PTSD
* current moderate or severe alcohol/drug use disorder or in the past 8 weeks
* current or past diagnosis of bipolar and other related disorders, schizophrenia spectrum, or other psychotic disorders
* concomitant treatments with medication known to have drug interactions with dronabinol, such as, central nervous system depressants (barbiturates, benzodiazepines, buspirone, lithium, etc) and anticholinergic agents (atropine, scopolamine, antihistamines, etc).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Rabinak, PhD, Principal Investigator — Wayne State University
Locations (1):
- Eugene Applebaum College of Pharmacy and Health Sciences, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Oral Capsule: Trauma-exposed individuals that received a one-time oral dose of placebo.
- Dronabinol Cap 5 Milligrams (MG): Trauma-exposed individuals that received a one-time oral dose of 5mg dronabinol.
- Dronabinol Cap 10 Milligrams (MG): Trauma-exposed individuals that received a one-time oral dose of 10mg dronabinol.
Period: Overall Study
Arm/Group | Placebo Oral Capsule | Dronabinol Cap 5 Milligrams (MG) | Dronabinol Cap 10 Milligrams (MG)
Started | 14 | 17 | 15
Completed | 12 | 16 | 15
Not Completed | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Oral Capsule: Trauma-exposed individuals with PTSD that received a one-time oral dose of placebo.
- Dronabinol Cap 5 Milligrams (MG): Trauma-exposed individuals with PTSD that received a one-time oral dose of 5mg dronabinol.
- Dronabinol Cap 10 Milligrams (MG): Trauma-exposed individuals with PTSD that received a one-time oral dose of 10mg dronabinol.
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Capsule | Dronabinol Cap 5 Milligrams (MG) | Dronabinol Cap 10 Milligrams (MG) | Total
Number analyzed (Participants) | 14 | 17 | 15 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 4
  Between 18 and 65 years | 13 | 16 | 13 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.29 (10.22) | 25.59 (9.81) | 25.13 (6.63) | 25.63 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 12 | 38
  Male | 1 | 4 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 16 | 15 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 5 | 14
  White | 7 | 9 | 8 | 24
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 15 | 46
CAPS-5 [Mean (Standard Deviation); unit: scores on a scale] — Clinician Administered PTSD Scale for DSM 5 Total severity score: Sum of values on the instrument that falls on a scale 0-80. Higher numbers represent more severe PTSD symptoms
  scores on a scale | 35.71 (12.29) | 35.65 (10.25) | 35.60 (12.27) | 35.66 (11.30)
PCL-5 [Mean (Standard Deviation); unit: scores on a scale] — PTSD Checklist for DSM 5 Total Score: Sum of values on the instrument that falls on a scale 0-80. Higher numbers represent more severe PTSD symptoms
  scores on a scale | 39.29 (17.17) | 45.71 (15.56) | 46.40 (16.65) | 43.99 (16.35)

OUTCOME MEASURES:

1. Primary Outcome: Brain Measures
Description: Mean functional magnetic resonance imaging (fMRI) BOLD activation extracted from each region of interests [amygdala; ventromedial prefrontal cortex; hippocampus] for each stimulus type (CS+E, CS+U, CS-). The units of BOLD values are expressed as arbitrary units.
Time Frame: Brain measures are collected on Visit 3, 14 days from baseline (Visit 1), Visit 4, 15 days from baseline (Visit 1), and Visit 5, 21 days from baseline (Visit 1), for approximately 1.5 hours each day
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Placebo Oral Capsule: In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (5mg or 10mg) or placebo (PBO) approximately two hours prior to MR scanning and task performance in 78 patients with PTSD.
  One-third of the participants will receive 5mg dronabinol (n=26) , one-third of the participants will receive 10mg dronabinol (n=26), and the remaining one-third of the participants will receive placebo (n=26).
  Placebo Oral Capsule: Placebo is administered only once (approximately 120 min prior to MR scanning in Visit 3) by the oral route and contains only dextrose in opaque capsules.
- Dronabinol Cap 5 Milligrams (MG): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (5mg or 10mg) or placebo (PBO) approximately two hours prior to MR scanning and task performance in 78 patients with PTSD.
  One-third of the participants will receive 5mg dronabinol (n=26) , one-third of the participants will receive 10mg dronabinol (n=26), and the remaining one-third of the participants will receive placebo (n=26).
  Dronabinol Cap 5 milligrams (MG): Dronabinol (5mg) is administered only once (approximately 120 min prior to MR scanning in Visit 3) by the oral route and is placed in an opaque capsule with dextrose filler.
- Dronabinol Cap 10 Milligrams (MG): In a randomized, double-blind, placebo-controlled, between-subjects design, we will administer a one-time oral dose of dronabinol (5mg or 10mg) or placebo (PBO) approximately two hours prior to MR scanning and task performance in 78 patients with PTSD.
  One-third of the participants will receive 5mg dronabinol (n=26) , one-third of the participants will receive 10mg dronabinol (n=26), and the remaining one-third of the participants will receive placebo (n=26).
  Dronabinol Cap 10 milligrams (MG): Dronabinol (10mg) is administered only once (approximately 120 min prior to MR scanning in Visit 3) by the oral route and is placed in an opaque capsule with dextrose filler.
Arm/Group | Placebo Oral Capsule | Dronabinol Cap 5 Milligrams (MG) | Dronabinol Cap 10 Milligrams (MG)
Number analyzed (Participants) | 11 | 11 | 14
arbitrary units
  Extinction Learning CS+E Amygdala-Visit 3 | 0.039567327 (0.241268856) | 0.092173636 (0.327156274) | 0.149446357 (0.335179325)
  Extinction Learning CS+E Hippocampus-Visit 3 | -0.021618 (0.186131283) | 0.000147182 (0.135589364) | 0.0734664 (0.112658087)
  Extinction Learning CS+E vmPFC-Visit 3 | -0.100398455 (0.251500983) | -0.140956909 (0.199637856) | -0.014101643 (0.20111521)
  Extinction Learning CS- Amygdala-Visit 3 | 0.058886909 (0.204782961) | -0.006294273 (0.261622699) | 0.160143 (0.241651249)
  Extinction Learning CS- Hippocampus-Visit 3 | -0.059069435 (0.127779008) | -0.133546182 (0.107201148) | -0.022569714 (0.101622507)
  Extinction Learning CS- vmPFC-Visit 3 | -0.108475118 (0.164705482) | -0.144499545 (0.207477253) | -0.058264393 (0.166826016)
  Recall CS+E Amygdala-Visit 4 | 0.064068818 (0.126060842) | 0.05063 (0.246216857) | 0.021313529 (0.144489742)
  Recall CS+E Hippocampus-Visit 4 | -0.018730882 (0.105994504) | -0.009476018 (0.079625507) | -0.008622411 (0.061309342)
  Recall CS+E vmPFC-Visit 4 | -0.092562327 (0.12096037) | -0.046500136 (0.148710336) | -0.042297714 (0.131211376)
  Recall CS- Amygdala-Visit 4 | 0.023179891 (0.369129301) | -0.045574364 (0.217199197) | 0.084785971 (0.188667772)
  Recall CS- Hippocampus-Visit 4 | 0.016318864 (0.130857648) | -0.012782118 (0.074290578) | 0.021303429 (0.086215257)
  Recall CS- vmPFC-Visit 4 | -0.025044173 (0.087226891) | -0.111483273 (0.136683884) | -0.023582643 (0.092589989)
  Recall CS+U Amygdala-Visit 4 | 0.073318518 (0.176984276) | -0.002491309 (0.192822633) | 0.106574214 (0.294631794)
  Recall CS+U Hippocampus-Visit 4 | 0.0027553 (0.114973037) | -0.048798436 (0.104668268) | 0.039578357 (0.157749137)
  Recall CS+U vmPFC-Visit 4 | -0.063881291 (0.195166763) | -0.11082 (0.125147494) | -0.068200429 (0.173367568)
  Renewal CS+E Amygdala-Visit 4 | -0.007166727 (0.16281838) | 0.085493291 (0.195124774) | -0.038971376 (0.225437092)
  Renewal CS+E Hippocampus-Visit 4 | -0.042572273 (0.121258736) | 0.053855418 (0.10101509) | 0.022821236 (0.09697586)
  Renewal CS+E vmPFC-Visit 4 | -0.025462455 (0.061109422) | -0.051927636 (0.137163274) | -0.044782714 (0.149704378)
  Renewal CS- Amygdala-Visit 4 | 0.038667909 (0.313060636) | 0.041082273 (0.249335278) | 0.089871571 (0.284506548)
  Renewal CS- Hippocampus-Visit 4 | 0.010737545 (0.135826418) | 0.028653909 (0.108329415) | 0.026597157 (0.177134712)
  Renewal CS- vmPFC-Visit 4 | -0.0115975 (0.174869566) | -0.035996455 (0.159479443) | 0.015976671 (0.173108329)
  Renewal CS+U Amygdala-Visit 4 | 0.033922182 (0.196452024) | -0.019035273 (0.347223043) | 0.04350675 (0.228228503)
  Renewal CS+U Hippocampus-Visit 4 | 0.001226509 (0.14949891) | 0.040038355 (0.128456906) | 0.037054743 (0.086797744)
  Renewal CS+U vmPFC-Visit 4 | -0.024311655 (0.109098602) | -0.063822713 (0.149376423) | -0.028642293 (0.086767322)
  Recall CS+E Amygdala-Visit 5 | 0.102081909 (0.267334482) | -0.112056636 (0.329023209) | 0.175857929 (0.2753103)
  Recall CS+E Hippocampus-Visit 5 | 0.066236364 (0.194500373) | -0.017467364 (0.172543206) | 0.127993357 (0.130790704)
  Recall CS+E vmPFC-Visit 5 | 0.0327043 (0.157330444) | -0.017208209 (0.168514694) | 0.007210571 (0.152128778)
  Recall CS- Amygdala-Visit 5 | 0.095167636 (0.307824688) | -0.060291409 (0.232370391) | 0.154838214 (0.250376068)
  Recall CS- Hippocampus-Visit 5 | 0.007481636 (0.231953032) | 0.006147773 (0.11636263) | 0.0426459 (0.145582746)
  Recall CS- vmPFC-Visit 5 | 0.017899909 (0.164153846) | -0.027662455 (0.149608896) | -0.056348421 (0.211452199)
  Recall CS+U Amygdala-Visit 5 | 0.067971218 (0.201754089) | 0.052176091 (0.407452643) | 0.089821286 (0.468006999)
  Recall CS+U Hippocampus-Visit 5 | 0.023053471 (0.152490758) | -0.009212182 (0.139630295) | 0.073768357 (0.26781902)
  Recall CS+U vmPFC-Visit 5 | -0.041723673 (0.105402346) | -0.024672805 (0.125923794) | -0.026101643 (0.16205021)
  Renewal CS+E Amygdala-Visit 5 | 0.061899727 (0.372039765) | 0.076936818 (0.234232725) | 0.091302143 (0.274868067)
  Renewal CS+E Hippocampus-Visit 5 | 0.063149555 (0.194680145) | 0.031223436 (0.165435695) | 0.031342243 (0.179872674)
  Renewal CS+E vmPFC-Visit 5 | 0.066609182 (0.266328372) | 0.040283 (0.147068638) | 0.048598129 (0.198056416)
  Renewal CS- Amygdala-Visit 5 | 0.183916727 (0.306917185) | 0.124069727 (0.211486836) | 0.15168205 (0.351211445)
  Renewal Hippocampus-Visit 5 | 0.013174 (0.209268027) | 0.056026436 (0.151187117) | 0.041636779 (0.19943295)
  Renewal CS- vmPFC-Visit 5 | 0.018359999 (0.217672587) | 0.0344149 (0.167694371) | -0.048354143 (0.323141034)
  Renewal CS+U Amygdala-Visit 5 | 0.312260455 (0.25005898) | 0.182693845 (0.255384016) | 0.095871914 (0.542394387)
  Renewal CS+U Hippocampus-Visit 5 | 0.111670727 (0.190179528) | 0.057369273 (0.133003425) | 0.009984107 (0.265241884)
  Renewal CS+U vmPFC-Visit 5 | 0.056020818 (0.195016729) | 0.085382818 (0.121708322) | 0.016284214 (0.334969996)
Statistical Analysis 1: Comparison: Placebo Oral Capsule vs Dronabinol Cap 5 Milligrams (MG) vs Dronabinol Cap 10 Milligrams (MG); Test type: Superiority; p < 0.05, ANOVA

2. Primary Outcome: Expectancy Ratings
Description: To assess the expected likelihood that an aversive cue (e.g. noise burst) will occur or not based on the CS shown on the screen. Participants rate their expectancy of the aversive cue using a button box on a scale from 1 to 3 [1 = certain that the aversive cue will be presented (Yes); 2 = certain that the aversive cue will not be presented (No); 3 = uncertain whether the aversive cue will be presented (I don't know)]. Counts of "yes", "no", and "I don't know" are collected on the first (early) trial of the CS and the last (late) trial of the CS.
Time Frame: Collected on Visit 2, 7 days from baseline (Visit 1), Visit 3, 14 days from baseline (Visit 1), Visit 4, 15 days from baseline (Visit 1), and Visit 5, 21 days from baseline (Visit 1) during the task. Each day the task lasts approximately 20 minutes.
Population: The number analyzed per row may differ from the overall analyzed due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Oral Capsule | Dronabinol Cap 5 Milligrams (MG) | Dronabinol Cap 10 Milligrams (MG)
Number analyzed (Participants) | 11 | 11 | 14
Participants
  Acquisition CS+E Early-Visit 2: number analyzed (Participants) | 11 | 10 | 12
  Acquisition CS+E Early-Visit 2: No | 3 | 5 | 4
  Acquisition CS+E Early-Visit 2: I Don't Know | 0 | 0 | 0
  Acquisition CS+E Early-Visit 2: Yes | 8 | 5 | 8
  Acquisition CS+U Early-Visit 2: number analyzed (Participants) | 11 | 10 | 12
  Acquisition CS+U Early-Visit 2: No | 0 | 2 | 2
  Acquisition CS+U Early-Visit 2: I Don't Know | 1 | 0 | 3
  Acquisition CS+U Early-Visit 2: Yes | 10 | 8 | 7
  Acquisition CS- Early-Visit 2: number analyzed (Participants) | 10 | 10 | 12
  Acquisition CS- Early-Visit 2: No | 6 | 9 | 5
  Acquisition CS- Early-Visit 2: I Don't Know | 1 | 0 | 3
  Acquisition CS- Early-Visit 2: Yes | 3 | 1 | 4
  Acquisition CS+E Late-Visit 2: number analyzed (Participants) | 10 | 10 | 13
  Acquisition CS+E Late-Visit 2: No | 2 | 2 | 6
  Acquisition CS+E Late-Visit 2: I Don't Know | 2 | 1 | 3
  Acquisition CS+E Late-Visit 2: Yes | 6 | 7 | 4
  Acquisition CS+U Late-Visit 2: number analyzed (Participants) | 11 | 10 | 13
  Acquisition CS+U Late-Visit 2: No | 3 | 4 | 1
  Acquisition CS+U Late-Visit 2: I Don't Know | 1 | 0 | 4
  Acquisition CS+U Late-Visit 2: Yes | 7 | 6 | 8
  Acquisition CS- Late-Visit 2: number analyzed (Participants) | 11 | 10 | 13
  Acquisition CS- Late-Visit 2: No | 11 | 7 | 9
  Acquisition CS- Late-Visit 2: I Don't Know | 0 | 0 | 1
  Acquisition CS- Late-Visit 2: Yes | 0 | 3 | 3
  Extinction CS+E Early-Visit 3: number analyzed (Participants) | 11 | 10 | 12
  Extinction CS+E Early-Visit 3: No | 2 | 1 | 4
  Extinction CS+E Early-Visit 3: I Don't Know | 1 | 4 | 4
  Extinction CS+E Early-Visit 3: Yes | 8 | 5 | 4
  Extinction CS- Early-Visit 3: number analyzed (Participants) | 10 | 10 | 13
  Extinction CS- Early-Visit 3: No | 4 | 3 | 4
  Extinction CS- Early-Visit 3: I Don't Know | 2 | 1 | 6
  Extinction CS- Early-Visit 3: Yes | 4 | 6 | 3
  Extinction CS+E Late-Visit 3: number analyzed (Participants) | 10 | 10 | 12
  Extinction CS+E Late-Visit 3: No | 9 | 9 | 9
  Extinction CS+E Late-Visit 3: I Don't Know | 0 | 1 | 2
  Extinction CS+E Late-Visit 3: Yes | 1 | 0 | 1
  Extinction CS- Late-Visit 3: number analyzed (Participants) | 11 | 10 | 13
  Extinction CS- Late-Visit 3: No | 11 | 9 | 9
  Extinction CS- Late-Visit 3: I Don't Know | 0 | 1 | 3
  Extinction CS- Late-Visit 3: Yes | 0 | 0 | 1
  Recall CS+E Early-Visit 4: number analyzed (Participants) | 11 | 9 | 13
  Recall CS+E Early-Visit 4: No | 4 | 7 | 9
  Recall CS+E Early-Visit 4: I Don't Know | 2 | 2 | 4
  Recall CS+E Early-Visit 4: Yes | 5 | 0 | 0
  Recall CS+U Early-Visit 4: number analyzed (Participants) | 11 | 9 | 13
  Recall CS+U Early-Visit 4: No | 3 | 7 | 3
  Recall CS+U Early-Visit 4: I Don't Know | 4 | 0 | 7
  Recall CS+U Early-Visit 4: Yes | 4 | 2 | 3
  Recall CS- Early-Visit 4: number analyzed (Participants) | 11 | 9 | 13
  Recall CS- Early-Visit 4: No | 8 | 6 | 7
  Recall CS- Early-Visit 4: I Don't Know | 2 | 3 | 5
  Recall CS- Early-Visit 4: Yes | 1 | 0 | 1
  Recall CS+E Late-Visit 4: number analyzed (Participants) | 11 | 10 | 14
  Recall CS+E Late-Visit 4: No | 11 | 9 | 11
  Recall CS+E Late-Visit 4: I Don't Know | 0 | 1 | 3
  Recall CS+E Late-Visit 4: Yes | 0 | 0 | 0
  Recall CS+U Late-Visit 4: number analyzed (Participants) | 10 | 11 | 14
  Recall CS+U Late-Visit 4: No | 10 | 10 | 11
  Recall CS+U Late-Visit 4: I Don't Know | 0 | 1 | 3
  Recall CS+U Late-Visit 4: Yes | 0 | 0 | 0
  Recall CS- Late-Visit 4: number analyzed (Participants) | 11 | 10 | 13
  Recall CS- Late-Visit 4: No | 11 | 9 | 10
  Recall CS- Late-Visit 4: I Don't Know | 0 | 1 | 3
  Recall CS- Late-Visit 4: Yes | 0 | 0 | 0
  Renewal CS+E Early-Visit 4: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS+E Early-Visit 4: No | 3 | 8 | 7
  Renewal CS+E Early-Visit 4: I Don't Know | 2 | 2 | 4
  Renewal CS+E Early-Visit 4: Yes | 6 | 1 | 2
  Renewal CS+U Early-Visit 4: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS+U Early-Visit 4: No | 5 | 8 | 7
  Renewal CS+U Early-Visit 4: I Don't Know | 3 | 2 | 5
  Renewal CS+U Early-Visit 4: Yes | 3 | 1 | 1
  Renewal CS- Early-Visit 4: No | 9 | 6 | 8
  Renewal CS- Early-Visit 4: I Don't Know | 2 | 2 | 6
  Renewal CS- Early-Visit 4: Yes | 0 | 3 | 0
  Renewal CS+E Late-Visit 4: number analyzed (Participants) | 10 | 10 | 13
  Renewal CS+E Late-Visit 4: No | 10 | 9 | 10
  Renewal CS+E Late-Visit 4: I Don't Know | 0 | 1 | 3
  Renewal CS+E Late-Visit 4: Yes | 0 | 0 | 0
  Renewal CS+U Late-Visit 4: number analyzed (Participants) | 10 | 10 | 14
  Renewal CS+U Late-Visit 4: No | 10 | 9 | 11
  Renewal CS+U Late-Visit 4: I Don't Know | 0 | 1 | 3
  Renewal CS+U Late-Visit 4: Yes | 0 | 0 | 0
  Renewal CS- Late-Visit 4: number analyzed (Participants) | 11 | 10 | 14
  Renewal CS- Late-Visit 4: No | 11 | 9 | 11
  Renewal CS- Late-Visit 4: I Don't Know | 0 | 1 | 3
  Renewal CS- Late-Visit 4: Yes | 0 | 0 | 0
  Recall CS+E Early-Visit 5: number analyzed (Participants) | 10 | 11 | 14
  Recall CS+E Early-Visit 5: No | 6 | 9 | 7
  Recall CS+E Early-Visit 5: I Don't Know | 3 | 2 | 6
  Recall CS+E Early-Visit 5: Yes | 1 | 0 | 1
  Recall CS+U Early-Visit 5: No | 7 | 9 | 8
  Recall CS+U Early-Visit 5: I Don't Know | 2 | 2 | 5
  Recall CS+U Early-Visit 5: Yes | 2 | 0 | 1
  Recall CS- Early-Visit 5: number analyzed (Participants) | 10 | 11 | 14
  Recall CS- Early-Visit 5: No | 5 | 8 | 6
  Recall CS- Early-Visit 5: I Don't Know | 2 | 2 | 6
  Recall CS- Early-Visit 5: Yes | 3 | 1 | 2
  Recall CS+E Late-Visit 5: number analyzed (Participants) | 10 | 11 | 14
  Recall CS+E Late-Visit 5: No | 10 | 10 | 10
  Recall CS+E Late-Visit 5: I Don't Know | 0 | 1 | 3
  Recall CS+E Late-Visit 5: Yes | 0 | 0 | 1
  Recall CS+U Late-Visit 5: number analyzed (Participants) | 10 | 10 | 14
  Recall CS+U Late-Visit 5: No | 10 | 9 | 10
  Recall CS+U Late-Visit 5: I Don't Know | 0 | 1 | 3
  Recall CS+U Late-Visit 5: Yes | 0 | 0 | 1
  Recall CS- Late-Visit 5: number analyzed (Participants) | 10 | 10 | 14
  Recall CS- Late-Visit 5: No | 10 | 9 | 10
  Recall CS- Late-Visit 5: I Don't Know | 0 | 1 | 3
  Recall CS- Late-Visit 5: Yes | 0 | 0 | 1
  Renewal CS+E Early-Visit 5: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS+E Early-Visit 5: No | 7 | 9 | 7
  Renewal CS+E Early-Visit 5: I Don't Know | 1 | 2 | 5
  Renewal CS+E Early-Visit 5: Yes | 3 | 0 | 1
  Renewal CS+U Early-Visit 5: number analyzed (Participants) | 11 | 11 | 12
  Renewal CS+U Early-Visit 5: No | 11 | 9 | 8
  Renewal CS+U Early-Visit 5: I Don't Know | 0 | 2 | 3
  Renewal CS+U Early-Visit 5: Yes | 0 | 0 | 1
  Renewal CS- Early-Visit 5: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS- Early-Visit 5: No | 9 | 8 | 7
  Renewal CS- Early-Visit 5: I Don't Know | 2 | 2 | 6
  Renewal CS- Early-Visit 5: Yes | 0 | 1 | 0
  Renewal CS+E Late-Visit 5: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS+E Late-Visit 5: No | 11 | 10 | 11
  Renewal CS+E Late-Visit 5: I Don't Know | 0 | 1 | 2
  Renewal CS+E Late-Visit 5: Yes | 0 | 0 | 0
  Renewal CS+U Late-Visit 5: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS+U Late-Visit 5: No | 11 | 10 | 11
  Renewal CS+U Late-Visit 5: I Don't Know | 0 | 1 | 2
  Renewal CS+U Late-Visit 5: Yes | 0 | 0 | 0
  Renewal CS- Late-Visit 5: number analyzed (Participants) | 11 | 11 | 13
  Renewal CS- Late-Visit 5: No | 11 | 10 | 10
  Renewal CS- Late-Visit 5: I Don't Know | 0 | 1 | 3
  Renewal CS- Late-Visit 5: Yes | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo Oral Capsule vs Dronabinol Cap 5 Milligrams (MG) vs Dronabinol Cap 10 Milligrams (MG); Test type: Superiority; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events are collected when a participant in enrolled in the study until study completion, which is approximately over a 3 week duration.
Arm/Group | Placebo Oral Capsule | Dronabinol Cap 5 Milligrams (MG) | Dronabinol Cap 10 Milligrams (MG)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/13 | 2/16 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Oral Capsule (N=13) | Dronabinol Cap 5 Milligrams (MG) (N=16) | Dronabinol Cap 10 Milligrams (MG) (N=15)
Nausea and Dizziness (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT03008005/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT03008005/ICF_001.pdf